CLINICAL TRIAL: NCT00847340
Title: Prevalence of HPV Genotypes in Genital Warts in Colombian Male and Female Population Attending Medical Services.
Brief Title: Human Papillomavirus (HPV) Genotypes in Genital Warts in Colombian Population
Acronym: GWprofamilia
Status: Completed | Type: Observational
Sponsor: La Fundacion para la Investigacion y el Desarrollo (Other)
Responsible Party: Principal Investigator, Gustavo Hernandez-Suarez, MD MSc, La Fundacion para la Investigacion y el Desarrollo
Other Study IDs: protocol V profamilia
Record Dates: First submitted 2009-02-17; First posted 2009-02-19 (Estimated); Last update posted 2012-03-20 (Estimated); Status verified 2012-03

CONDITIONS: Genital Warts; HPV Infections
Keywords: Genital warts; HPV typing; HPV infections; Condyloma Acuminata
MeSH Terms: conditions — Condylomata Acuminata; Papillomavirus Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Biopsies from genital warts will be taken through an excisional procedure. Homeostasis will be obtained by using topications of Monssell solution. Biopsy sample will be splinted in order to obtain two pieces, one of them will be frozen (liquid Nitrogen) and designated to the HPV DNA PCR test (GP5, GP6) to be performed at the immunology lab at the National Cancer Institute in Bogotá. The other one will be kept in Formalin solution (10%) and sent to the pathology laboratory for haematoxiline - eosine paint and lecture.
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Biopsy Excisional — Biopsied from genital warts will be taken through an excisional procedure. Homeostasis will be obtained by using apply of Monsel solution. Biopsied sample will be splinted in order to obtain two pieces, one of them will be frozen (liquid Nitrogen) and designated to the HPV DNA PCR test (GP5, GP6) to be performed at the immunology lab at the National Cancer Institute in Bogotá. The other one will be kept in Formalin solution (10%) and sent to the pathology laboratory for haematoxiline - eosine paint and lecture.
  Other Names: Resection genital warts

SUMMARY:
HPV infection has been recognized as the most prevalent sexual transmitted infection worldwide. Burden of many HPV related diseases is well known particularly regarding the different associated cancers (cervical, anal, vaginal, vulvar, oro-pharyngeal) (3) ; however, there is much less available information on the general burden of genital warts, the associated HPV types, the costs of related medical treatments and the knowledge and perceptions towards the disease and its prevention.

Objectives:

1. To determine the HPV genotypes distribution in genital warts in the study population.
2. To assess the knowledge about transmission & prevention of HPV infection related diseases
3. To determine the direct medical costs of genital warts attention.

DETAILED DESCRIPTION:
Study population

Female and male between 18 - 45 years of age living in Bogota, Colombia

Sample frame

Patients attending to gynecologic or STD consult in a mayor out patient clinic in Bogotá (PROFAMILIA)

Analysis

Analysis of the information will be exhaustive. We will calculate prevalence of HPV genotypes in the GW in both sexes separately. Analyses of the survey will include simple frequencies, percentages, and comparison of results related to HPV knowledge with sociodemographic and clinical information. Explorative analysis using parametric or non parametric statistics of the items included in the questionnaire and clinical forms will be done as appropriate. We will calculate the medical cost of patients enrolled in the study. The treatment protocols used for this protocol will reflect the current clinical practice accepted for the treatment of genital warts. We will use national reference cost list (SOAT) to determine the cost of procedures included.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-45 years.
* Lesions suspicious of being HPV related.
* The main manifestations of anogenital warts include:

  * Cauliflower-like condylomata acuminata lesions that usually involve moist surfaces
  * keratotic and smooth papular warts, usually on dry surfaces
  * subclinical "flat" warts, that can be found on any mucosal or cutaneous surface and, which are probably overseen in the majority of cases.
* Lesions other than the described above, are not to be biopsied, according to the investigator criteria.

Exclusion Criteria:

* Not willing to participate
* To be a participant in any HPV vaccine clinical trial study
* Known immune suppressive disease.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients attending to gynecologic or STD consult in a mayor out patient clinic in Bogotá (PROFAMILIA).
  Female and male between 18 - 45 years of age living in Bogota, Colombia.
Sampling Method: Non-Probability Sample
Enrollment: 342 (Actual)
Dates: Start 2009-12; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gustavo J. Hernandez-Suarez, MD, Principal Investigator — Research & Development Fundation (FID)